CLINICAL TRIAL: NCT01725594
Title: A Two-Part, Phase 1, Single and Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of CAT-2003 in Healthy Subjects
Brief Title: A Single and Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of CAT-2003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CAT-2003-101
Record Dates: First submitted 2012-11-06; First posted 2012-11-14 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Cohort A1, Dose Level 1: CAT 2003 or placebo fasting (Experimental): Single dose
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort A2, Dose Level 2: CAT 2003 or placebo fasting (Experimental): Single dose
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort A3, Dose Level 3: CAT 2003 or placebo fasting (Experimental): Single dose
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort A4, Dose Level 4: CAT 2003 or placebo fasting (Experimental): Single dose
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort A5, Dose Level 5: CAT 2003 or placebo fasting (Experimental): Single dose
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort A2: Dose Level 2: CAT 2003 or placebo fed (Experimental): Single dose
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort A3: Dose level 3:CAT 2003 or placebo fed (Experimental): Single dose
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort B1: Dose level 6: CAT 2003 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort B2: Dose level 7: CAT 2003 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort B3: Dose level 8: CAT 2003 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT 2003; Drug: Placebo
- Cohort B4: Dose level 9: CAT 2003 or placebo (Experimental): Multiple dose for 14 days
  Interventions: Drug: CAT 2003; Drug: Placebo

INTERVENTIONS:
Drug: CAT 2003
Drug: Placebo

SUMMARY:
This is a two-part Phase 1 placebo-controlled, double-blind, randomized single and multiple ascending dose study. In Part A, CAT-2003 is administered as a single dose; at two doses (1000 and 2000 mg), subjects will return for a second dose of CAT-2003 or placebo after a high fat meal. In Part B, CAT-2003 is administered for 14 consecutive days.

ELIGIBILITY:
Major Inclusion Criteria:

* Provision of written informed consent prior to any study-specific procedure;
* Good health as determined by medical history, physical examination, vital signs, ECG, and clinical laboratory measurements;
* Satisfies one of the following:

  1. Females not of childbearing potential: non-pregnant and non-lactating; surgically sterile or postmenopausal for 2 years or at least 1 year with a follicle stimulating hormone assessment (FSH) greater than or equal to 40 IU/L; OR
  2. Males: surgically sterile, abstinent, or subject or partner is utilizing an acceptable contraceptive method during and 3 months after the last study dose;

Major Exclusion Criteria:

* Clinically significant disease that requires a physician's care and/or would interfere with study evaluations
* Clinically significant electrocardiogram (ECG) abnormalities or laboratory results as assessed by the investigator, such as QTcF >450;
* Use of any investigational drug or participation in any investigational study within 30 days prior to screening or 5 half-lives of the study agent, whichever is longer;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | Screening to End of study (up to 4 weeks following randomization)

SECONDARY OUTCOMES:
AUCinf of CAT-2003 | Days 1, 7 and 14
Cmax of CAT-1004 | Days 1, 7 and14
Changes from baseline for hematology, chemistry, coagulation and urinalysis | Baseline through End of study (up to 4 weeks)
Changes from baseline for Physical exams | Baseline through end of study (up to 4 weeks)
Changes from baseline for ECGs | Baseline through end of study (up to 4 weeks)
Changes from baseline in vital signs | Baseline through end of study (up to 4 weeks)
Assess the pharmacodynamic effects of multiple doses of CAT-2003 on triglycerides and other lipids (LDL-C, VLDL-C, VLDL-triglycerides, non-HDL-C, total cholesterol, HDL-C), apoB, lipoprotein(a), and PCSK9 in healthy subjects with mild dyslipidemia | Baseline to end of study (up to 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Biernat, M.D, Principal Investigator — Medpace, Inc.
Locations (1):
- Medpace CPU, Cincinnati, Ohio, United States